CLINICAL TRIAL: NCT04864912
Title: A Retrospective Mapping of Health Care Utilisation and Current Quality of Life Status in Adult Subjects With a History of Chronic Otitis Media With or Without Cholesteatoma Who Have Undergone a Primary Tympanoplasty
Brief Title: Retrospective Health Care Utilisation and Current Quality of Life in Adults With Chronic Otitis Media Who Had a Middle Ear Surgery
Status: Completed | Type: Observational
Sponsor: Cochlear (Industry)
Collaborators: QbD Clinical (Industry); Suministros Hospitalarios Medical Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: CBAS5780
Record Dates: First submitted 2021-04-13; First posted 2021-04-29 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Chronic Otitis Media
Keywords: Primary tympanoplasty
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires and survey — Questionnaires: Health Utilities Index Mark III, Chronic Otitis Media Outcome Test-15 and Speech, Spatial, and Qualities of Hearing Scale-12 Survey: Client Service Receipt Inventory (adapted version)

SUMMARY:
The objective of this multicentre study is to evaluate the standard of care of participants diagnosed with Chronic Otitis Media that have already gone through a first middle ear surgery but still have at least a moderate hearing loss. The study has a retrospective part (extraction of medical chart data) and a prospective part with a survey and three questionnaires collecting data on the use of health care services, on health related quality of life and hearing performance.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, 18 years or older.
* Subjects with conductive or mixed hearing loss.
* Subjects with historically documented diagnosis of Chronic Otitis Media (COM) with or without cholesteatoma in the operated ear.
* Subjects who have undergone primary tympanoplasty type I-V to improve hearing between 2010-2016.
* Subjects with a Pure Tone Average (PTA)4 air-bone gap ≥30 decibels (dB) OR PTA4 air-bone gap between 25-30 dB with an air conduction threshold PTA4 ≥40 dB HL within 12 months after primary tympanoplasty in the operated ear.
* Subjects who have been recommended by their health care professional to try a hearing aid to improve hearing in the operated ear.
* Pre-op audiogram, maximum 1 year prior to the primary tympanoplasty, and post-op audiogram for the primary tympanoplasty are available.
* Aided audiogram, unaided if no hearing device is used, available between 2018 and the point of enrolment.
* Subjects are fluent in the language used for study questionnaires: German, French, Spanish.
* Subjects are willing and able to provide written informed consent. For France: subjects do not oppose to participate in the study.
* Medical Record data is available throughout the defined data search period, from primary tympanoplasty to point of enrolment.

Exclusion Criteria:

* Subjects are unable or unwilling to comply with the requirements of the study as determined by the investigator.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this study.

For France only:

* Subjects who are not affiliated to social security.
* Subjects who are under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with a history of chronic otitis media who have undergone a primary tympanoplasty to improve hearing between 2010-2016 but still have conductive or mixed hearing loss.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christiane D'hondt, Study Director — Cochlear
Locations (6):
- France (2):
  - Hôpital Bicêtre, Hôpitaux universitaires Paris Sud AP-HP, Le Kremlin-Bicêtre
  - ENT department - Bâtiment Pierre Paul Riquet - Hôpital Purpan, Toulouse
- Germany (2):
  - Universitätsklinik für Hals-, Nasen und Ohrenheilkunde, Freiburg im Breisgau
  - Hals-, Nasen- und Ohrenklinik, Universitätsklinikum Heidelberg, Heidelberg
- Spain (2):
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational Cohort: Adult participants with a history of chronic otitis media who have undergone a primary tympanoplasty to improve hearing between 2010-2016 but still have conductive or mixed hearing loss.
Period: Overall Study
Arm/Group | Observational Cohort
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Observational Cohort
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (18.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diabetes [Number; unit: participants]
  No | 65
  Yes | 4
Turner Syndrome [Number; unit: participants]
  No | 69
  Yes | 0
Cleft Palate [Number; unit: participants]
  No | 69
  Yes | 0
Down Syndrome [Number; unit: participants]
  No | 69
  Yes | 0
Cholesteatoma [Number; unit: participants]
  No | 33
  Yes | 36

OUTCOME MEASURES:

1. Primary Outcome: Number and Type of Contacts With Health Care Providers
Description: Contacts are obtained from medical records, counted and categorized.
Time Frame: From primary tympanoplasty to time of enrolment, up to 13 years
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Cohort
Number analyzed (Participants) | 69
Participants
  Contact for 1 surgical procedure | 45
  Contact for 2 surgical procedures | 14
  Contact for 3 surgical procedures | 5
  Contact for 4 surgical procedures | 3
  Contact for more than four surgical procedures | 2
  Contact for 2 audiograms | 45
  Contact for 3 audiograms | 5
  Contact for 4 audiograms | 3
  Contact for more than four audiograms | 16
  1 other healthcare contacts | 5
  2 other healthcare contacts | 1
  3 other healthcare contacts | 4
  4 other healthcare contacts | 7
  More than 4 other healthcare contacts | 36

2. Primary Outcome: Number and Type of Interventions and/or Procedures
Description: Medical examinations, surgical procedures and hearing rehabilitation are obtained from medical records, counted and categorized.
Time Frame: From primary tympanoplasty to time of enrolment, up to 13 years
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Cohort
Number analyzed (Participants) | 69
Participants
  CT scan of the temporal bone and/or sinuses | 12
  MRI of the temporal bone or the brain | 23
  another medical examination | 14
  primary tympanoplasty | 65
  revision surgeries | 25
  planned staged or second look surgeries | 18

3. Primary Outcome: Number and Type of Medications and Therapies
Description: Medications are obtained from medical records, counted and categorized. Therapies from medical records are listed.
Time Frame: From primary tympanoplasty to time of enrolment, up to 13 years
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Cohort
Number analyzed (Participants) | 69
Participants
  Antiinfective | 20
  Analgesics and anesthetics | 1
  Anilides | 14
  Antivertigo preparations | 3
  Benzodiazepine derivatives | 1
  Combinations of penicillins, incl. beta-lactamase inhibitors | 4
  Corticosteroids | 5
  Corticosteroids and antiinfectives in combination | 12
  Fluoroquinolones | 3
  Glucocorticoids | 5
  Macrolides | 1
  Other otologicals | 2
  Other cicatrizants | 1
  Other opioids | 6
  Penicillins with extended spectrum | 2
  Pyrazolones | 2

4. Secondary Outcome: Hearing Performance Assessed Via an Audiogram
Description: PTA4 (0.5, 1, 2 and 4 kHz) for both air and bone conduction, under unaided and when applicable aided conditions. Data obtained from participant medical records.
Time Frame: Up to 12 months prior to primary tympanoplasty
Population: Bone conduction studies were not carried out for all participants
Measure: Mean (Standard Deviation); unit: db HL (decibel hearing loss)
Arm/Group | Observational Cohort
Number analyzed (Participants) | 69
db HL (decibel hearing loss)
  Air Conduction | 53.2 (19.64)
  Bone Conduction: number analyzed (Participants) | 42
  Bone Conduction | 23.8 (14.76)

5. Secondary Outcome: Hearing Performance Assessed Via an Audiogram
Description: as for outcome 4
Time Frame: Within 12 months after primary tympanoplasty
Population: Bone conduction studies were not carried out for all participants
Measure: Mean (Standard Deviation); unit: db HL (decibel hearing loss)
Arm/Group | Observational Cohort
Number analyzed (Participants) | 69
db HL (decibel hearing loss)
  Air Conduction | 58.7 (14.9)
  Bone conduction: number analyzed (Participants) | 37
  Bone conduction | 25.3 (14.85)

6. Secondary Outcome: Hearing Performance Assessed Via an Audiogram
Description: as for outcome 4
Time Frame: Up to 6 years prior to study enrollment
Population: Bone conduction studies were not carried out for all participants
Measure: Mean (Standard Deviation); unit: db HL (decibel hearing loss)
Arm/Group | Observational Cohort
Number analyzed (Participants) | 69
db HL (decibel hearing loss)
  Air conduction: number analyzed (Participants) | 68
  Air conduction | 56.7 (21.16)
  Bone conduction: number analyzed (Participants) | 31
  Bone conduction | 25.2 (13.89)

7. Secondary Outcome: Health Care Costs
Description: Direct medical costs were calculated by applying the reported Diagnosis Related Group (DRG) codes for Chronic Otitis Media related health care utilization were obtained to the unit cost in each participating country for each participant.
  Note: No outcome measures are reported as there was insufficient data collection
Time Frame: From primary tympanoplasty to time of enrolment.
Population: A small number of DRG codes from only a single clinic were reported in this study. A cost could not be directly linked to these codes as the hospitals negotiate the tariffs with the health insurers and these tariffs are not made public. Hence, despite having collected a small number of codes, the health care costs could not be calculated, and results are not available for this outcome measure.
Arm/Group | Observational Cohort
Number analyzed (Participants) | 0

8. Secondary Outcome: Socio-economic Status and Health Care Data Via the Client Service Receipt Inventory (CSRI) Survey
Description: Demographic data, medical history, hearing rehabilitation, health care utilisation related to ear infection and hearing difficulties and employment information data are collected.
Time Frame: At enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Cohort
Number analyzed (Participants) | 69
Participants
  married/living as married | 41
  single | 14
  widowed | 7
  divorced/separated | 6
  living with spouse/partner and children | 24
  living with spouse/partner without children | 19
  living alone | 13
  living with their parents | 6
  lived in other conditions | 6
  place of residence was an owner occupied flat/house | 44
  place of residence was a privately rented flat/house | 15
  place of residence was a flat/house rented from a local authority or housing association | 4
  other places of residence | 5
  highest level of education was university or higher | 20
  highest level of education was high school | 19
  highest level of education was vocational training | 17
  highest level of education was primary school | 12
  high blood pressure | 12
  autoimmune disease | 4
  cancer | 1
  heart disease | 5
  diabetes | 4
  chronic lung disease | 4
  chronic kidney disease | 2
  mood disorders | 8
  substance dependency | 1
  other chronic disease | 13
  never smoked | 39
  current smokers | 16
  previous smokers | 13
  full-time employment | 31
  retired | 20
  part-time employment | 5
  retired (because of ill health), unemployed, student or housewife/husband | 2
  self-employed | 1
  currently use a hearing aid or hearing device | 31
  bone conduction implant | 7
  visited a general practitioner | 21
  attended a day hospital or accident and emergency | 2
  visited an ENT | 31
  Visited audiologist | 14

9. Secondary Outcome: Self-reported Health Status and Health Related Quality of Life Via the Health Utilities Index Mark III (HUI3) Questionnaire.
Description: HUI provides descriptive evidence on multiple dimensions of health status, a score for each dimension of health and an overall Health Related Quality of life score. The HUI3 classification system is comprised of 8 attributes: Vision, Hearing, Speech, Ambulation, Dexterity, Emotion, Cognition and Pain - each with 5 or 6 levels of ability/disability The scoring systems provide utility (preference) scores on a generic scale where 0.00 indicates death and 1.00 indicates perfect health.
Time Frame: At enrolment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Observational Cohort
Number analyzed (Participants) | 67
score on a scale
  Overall | 0.7 (0.28)
  Vision | 0.9 (0.17)
  Hearing | 0.8 (0.29)
  Speech | 0.9 (0.15)
  Dexterity | 1 (0.11)
  Emotion | 0.9 (0.16)
  Cognition | 0.9 (0.14)
  Pain | 0.9 (0.19)

10. Secondary Outcome: Self-reported Health Related Quality of Life of Participants With COM Via the Chronic Otitis Media Outcome Test-15 (COMOT-15) Questionnaire.
Description: COMOT-15 measures Health Related Quality of life of participants with COM. It consists of three subscales: ear symptoms, hearing function, and mental health forming the overall score. In addition, two questions related to COM are asked: one on the general evaluation of quality of life and one on the frequency of doctor visits in the last six months. The total score and the sub-scores are transformed to a 0-100 scale by dividing the sum of the raw scores of the items by the sum of spans of the items, then multiplying by 100. A higher score indicates a worse health-related quality of life.
Time Frame: At enrolment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Observational Cohort
Number analyzed (Participants) | 68
units on a scale
  Overall | 43 (18.25)
  Ear symptoms | 29.4 (20.28)
  Hearing function | 65 (22.84)
  Mental Health | 46.5 (27.31)

11. Secondary Outcome: Self-reported Auditory Disability Via the Speech, Spatial and Qualities of Hearing Scale (SSQ-12) Questionnaire
Description: SSQ-12 measures speech, spatial and hearing experiences. The total(overall) score summarizes these parameters. A scale from 0 to 10 is used. A mark 0 means "be quite unable to do or experience what is described" and a mark 10 means "be perfectly able to do or experience what is described in the question".
Time Frame: At enrolment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Observational Cohort
Number analyzed (Participants) | 65
score on a scale | 5.5 (2.18)

12. Secondary Outcome: Chronic Otitis Media Outcome Test -15 (COMOT-15) Questionnaire in German, French and Spanish
Description: Mean score of Chronic Otitis Media Outcome Test -15 (COMOT-15) in German, French and Spanish (0-100 scale). This questionnaire consists of 15 questions that query 3 subscales: ear symptoms, hearing function, and mental health. Additionally, it includes a question about quality of life and specialist doctor visit frequency.
  The total score is summed, transformed and presented on a 0 - 100 scale where 0 is a good outcome and 100 is the worst possible outcome.
Time Frame: At enrollment
Population: Participants only completed the questionnaire in one language and one participant in the study did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale (0-100)
Arm/Group | Observational Cohort
Number analyzed (Participants) | 68
score on a scale (0-100)
  German: number analyzed (Participants) | 19
  German | 36.8 (14.76)
  French: number analyzed (Participants) | 17
  French | 46.3 (22.73)
  Spanish: number analyzed (Participants) | 32
  Spanish | 45 (17.12)

ADVERSE EVENTS:
Time Frame: Not applicable. Survey administered at a single timepoint and retrospective chart review design.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed due to cross-sectional and retrospective chart review study design.
Arm/Group | Observational Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication would be a joint publication covering data from all centers, and subsequent publications will refer to that first publication. Investigators can publish or present after agreement between the Coordinating and Principal Investigators, and the Sponsor after the main publication is submitted and approved. Conference presentations or publications must be sent for review at least to the Sponsor 30 - 60 days (site-specific) prior to submission or presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT04864912/Prot_SAP_000.pdf